CLINICAL TRIAL: NCT07091695
Title: Real-world Outcomes Among Patients With Melanoma Treated With Neoadjuvant Nivolumab+Relatlimab (Nivo+Rela) or Nivolumab+Ipilimumab (Nivo+Ipi)
Brief Title: Real-world Outcomes Among Patients With Melanoma Treated With Neoadjuvant Nivolumab+Relatlimab or Nivolumab+Ipilimumab
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA224-1084
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; relatlimab; Ipilimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants receiving nivolumab + relatlimab treatment
  Interventions: Biological: Nivolumab + relatlimab
- Participants receiving nivolumab + ipilimumab treatment
  Interventions: Biological: Nivolumab + ipilimumab

INTERVENTIONS:
Biological: Nivolumab + relatlimab — As prescribed by the treating clinician
  Groups: Participants receiving nivolumab + relatlimab treatment
Biological: Nivolumab + ipilimumab — As prescribed by the treating clinician
  Groups: Participants receiving nivolumab + ipilimumab treatment

SUMMARY:
The purpose of this study is to understand the characteristics of adults diagnosed with with clinically palpable stage III resectable melanoma, the associated treatment patterns for their disease, and outcomes associated with the real-world use of neoadjuvant nivolumab+relatlimab or nivolumab+ipilimumab

ELIGIBILITY:
Inclusion Criteria:

* Participants at least 18 years old at diagnosis of clinically palpable stage III resectable melanoma
* Participants treated with nivolumab+relatimab (nivo+rela) or nivolumab+ipilimumab (nivo+ipi) in the neoadjuvant setting
* Participants with at least 6 months of follow-up from initiation of neoadjuvant therapy, unless deceased prior to 6 months of follow-up

Exclusion Criteria:

* Participants received nivo+rela or nivo+ipi for clinically palpable stage III resectable melanoma as part of a therapeutic clinical trial
* Participants had history of diagnosis of any malignancy (except for non-melanoma skin cancer) in the last 2 years.
* Participants received adjuvant nivo+rela or adjuvant nivo+ipi after neoadjuvant nivo+ipi
* Participants received adjuvant nivo+ipi after neoadjuvant nivo+rela
* Participants received any systemic therapy prior to the initiation of neoadjuvant nivo+rela or nivo+ipi

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise of adult diagnosed with clinically palpable stage III resectable melanoma in the U.S. managed by physicians in Cardinal Health's OPEN treated with neoadjuvant nivolumab+relatimab or nivolumab+ipilimumab from 18 March 2022.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-05-11 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Participant baseline demographics | Baseline
Participant baseline clinical characteristics | Baseline
Participant treatment history | Baseline
Number of doses of index therapies received (neoadjuvant therapies) | Day 1
Types of surgeries received for melanoma after the index date | Up to 42-months
Date of last radiation received for melanoma after the index date | Up to 42-months
Types of regimens received for melanoma post-surgery in the adjuvant setting | Up to 42-months
Number of doses of adjuvant therapies received (post-surgery) | Up to 42-months
Dose modifications received by participants | Up to 42-months
Rationale for dose modifications | Up to 42-months
Rationale for treatment discontinuation | Up to 42-months
Overall survival (OS) | Up to 42-months
Time to treatment discontinuation (TTD) | Up to 42-months
Duration of treatment (DOT) | Up to 42-months
Time from neoadjuvant index treatment to adjuvant therapy | Up to 42-months
Time from neoadjuvant index treatment to surgery | Up to 42-months
Time from surgery to adjuvant therapy | Up to 42-months
Pathologic complete response (PCR) | Up to 42-months
Event-free survival (EFS) | Up to 42-months
Distant metastasis-free survival (DMFS) | Up to 42-months
Participant adverse events (AEs) | Up to 42-months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Cardinal Health, Dublin, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts